CLINICAL TRIAL: NCT01013246
Title: Effects of Playing Video Games on Energy Balance: a Randomized, 2-condition, Crossover Study in Adolescents
Brief Title: Effects of Playing Video Games on Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Anders M. Sjödin, MD, PhD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B268
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
Keywords: Video games; Energy balance; Metabolism; Appetite control
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video game play (Experimental)
  Interventions: Other: 1-hour video game play

INTERVENTIONS:
Other: 1-hour video game play — FIFA 2009, a football video game played on Xbox 360

SUMMARY:
The aim of this study is to examine the effects of playing video games on various components of energy balance and substrate metabolism as well as on glucose homeostasis and relevant hormonal systems that might be involved in the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescents between 15 and 19 years of age
* Normal weight (5th percentile to less than the 85th percentile)

Exclusion Criteria:

* Smoking
* Unstable body weight (±4 kg) during the 6 months preceding testing
* Regular physical exercise (>3 hours/week)
* Excessive intake of alcohol (>7 drinks/week)
* Substance abuse
* Metabolic disease (e.g. thyroid disease, heart disease, diabetes, etc.)
* Medication that could interfere with the outcome variables
* Eating disorder
* High restraint eating behavior (score ≥8 for cognitive dietary restraint in the Three-Factor Eating Questionnaire)
* Irregular eating schedule (e.g. skipping breakfast)
* Unfamiliar with the use of video games
* Unable to comply with the protocol

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Energy intake and energy expenditure | 1 time point

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Chaput JP, Visby T, Nyby S, Klingenberg L, Gregersen NT, Tremblay A, Astrup A, Sjodin A. Video game playing increases food intake in adolescents: a randomized crossover study. Am J Clin Nutr. 2011 Jun;93(6):1196-203. doi: 10.3945/ajcn.110.008680. Epub 2011 Apr 13. PMID 21490141